CLINICAL TRIAL: NCT00424424
Title: Proprietary Information - Exploratory (Non-Confirmatory) Trial
Brief Title: A Study to Evaluate the Efficacy of MK0719 in the Prevention of Postoperative Dental Pain (0719-002)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 0719-002; 2007_505
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Pain, Postoperative
Keywords: Postoperative Dental Pain
MeSH Terms: conditions — Pain, Postoperative

INTERVENTIONS:
Drug: MK0719

SUMMARY:
This study is being conducted to evaluate the safety and tolerability of the drug and to evaluate its efficacy compared to placebo and to ibuprofen in the prevention of postoperative dental pain in male patients.

This is an early phase trial and some specific protocol information is proprietary and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria :

* Patients in generally good health who are scheduled to have 2 or more third molars removed, at least 1 of which is partially or completely embedded in bone and is a mandibular impaction

Exclusion Criteria :

* Patient has a history of any illness or condition that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2006-08; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Proprietary Information - Exploratory (Non-Confirmatory) Trial

SECONDARY OUTCOMES:
Proprietary Information - Exploratory (Non-Confirmatory) Trial

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC